CLINICAL TRIAL: NCT00718809
Title: Phase II Trial of AZD0530 for Patients With Relapsed/Refractory Thymic Malignancies (Thymoma and Thymic Carcinoma)
Brief Title: Saracatinib in Treating Patients With Relapsed or Refractory Thymoma or Thymic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00297; IUCRO-0214
Record Dates: First submitted 2008-07-18; First posted 2008-07-21 (Estimated); Results first posted 2015-06-10 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2014-10

CONDITIONS: Invasive Thymoma and Thymic Carcinoma; Recurrent Thymoma and Thymic Carcinoma; Stage III Thymoma; Stage IVA Thymoma; Stage IVB Thymoma
MeSH Terms: conditions — Thymoma | interventions — saracatinib

ARMS (1):
- Arm I (Experimental): Patients receive oral saracatinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: saracatinib

INTERVENTIONS:
Drug: saracatinib — Given orally
  Other Names: AZD0530

SUMMARY:
This phase II trial is studying how well saracatinib works in treating patients with relapsed or refractory thymoma or thymic cancer. Saracatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the objective response rate (complete response and partial response) in patients with relapsed or refractory thymoma or thymic carcinoma treated with AZD0530.

SECONDARY OBJECTIVES:

I. To evaluate the toxicity of AZD0530 in these patients. II. To evaluate the progression-free survival of these patients. III. To evaluate the overall survival of these patients. IV. To evaluate the disease control rate, defined as complete response, partial response, and stable disease, in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral saracatinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive thymoma or thymic carcinoma, meeting the following criteria:

  * Relapsed or refractory disease
  * Metastatic, unresectable disease
  * Locally invasive disease allowed provided it is not resectable and has been previously treated
  * Progressive disease
* Measurable disease, defined as >= 1 unidimensionally measurable lesion >= 20 mm by conventional techniques or >= 10 mm by spiral CT scan
* Must have received >= 1 prior chemotherapy regimen
* No active brain metastases
* Patients with previously treated brain metastases (surgical resection or radiotherapy) are eligible provided they have documented stable brain disease for >= 1 month after completion of therapy and are asymptomatic
* ECOG performance status 0-2
* Leukocytes >= 3,000/mm^3
* ANC >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin > 9 g/dL
* Serum bilirubin < 2.0 times upper limit of normal (ULN)
* Transaminases =< 2.5 times ULN (< 5.0 times ULN if liver metastasis is present)
* Serum creatinine < 1.5 times ULN OR creatinine clearance > 50 mL/min
* Urine protein:creatinine ratio < 0.5 OR urine protein < 1,000 mg by 24-hour urine collection
* QTc < 460 msec
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 30 days after completion of study treatment
* No known history of allergic reactions attributed to compounds of similar chemical or biological composition to AZD0530
* No other malignancies within the past 3 years, except curatively treated in situ carcinoma of the cervix or completely resected nonmelanoma skin cancer
* No concurrent active malignancies other than thymic malignancy
* No condition that impairs the ability to swallow AZD0350 tablets (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease)
* No cardiac dysfunction including, but not limited to, any of the following:

  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * History of ischemic heart disease
  * Myocardial infarction within the past year
  * No QTc prolongation or other significant ECG abnormalities
  * No poorly controlled hypertension (i.e., systolic blood pressure [BP] ≥ 150 mm Hg or diastolic BP ≥ 95 mm Hg)
* No evidence of severe or uncontrolled systemic conditions that would make it undesirable to participate in the study or that would jeopardize compliance with the study, including any of the following:

  * Severe hepatic impairment
  * Interstitial lung disease (bilateral, diffuse, or parenchymal lung disease)
  * Unstable or uncompensated respiratory condition
  * Unstable or uncompensated cardiac condition
* No uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Mental health issues or social circumstances that would limit compliance with study requirements
* No prior src inhibitors
* At least 4 weeks since prior systemic therapy (6 weeks for carmustine or mitomycin C)
* At least 8 weeks since prior immunotherapy
* At least 4 weeks since prior octreotide
* Concurrent octreotide for pure red cell aplasia allowed provided patient continues on the same dose and schedule, has had a response to this drug, and has demonstrated progressive thymoma by radiography or physical exam
* At least 4 weeks since prior surgery and recovered
* At least 4 weeks since prior investigational agents
* At least 4 weeks since prior radiotherapy to measurable disease sites (2 weeks for palliative radiotherapy to metastatic sites) and recovered
* At least 7 days since prior and no concurrent active CYP3A4 agents or substances
* No other concurrent investigational or anticancer agents
* No concurrent combination antiretroviral therapy for HIV-positive patients
* Concurrent steroids allowed for treatment of a pre-existing autoimmune disorder or as antiemetic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-06; Primary Completion 2010-08 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Loehrer, Principal Investigator — Indiana University School of Medicine
Locations (2):
- United States (2):
  - Stanford University Hospitals and Clinics, Stanford, California
  - Indiana University Medical Center, Indianapolis, Indiana

REFERENCES:
- [Derived] Gubens MA, Burns M, Perkins SM, Pedro-Salcedo MS, Althouse SK, Loehrer PJ, Wakelee HA. A phase II study of saracatinib (AZD0530), a Src inhibitor, administered orally daily to patients with advanced thymic malignancies. Lung Cancer. 2015 Jul;89(1):57-60. doi: 10.1016/j.lungcan.2015.04.008. Epub 2015 Apr 25. PMID 26009269

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This protocol was based on getting at least 12 eligible patients with thymoma to complete stage one. There are 12 eligible thymoma patients and also 9 thymic carcinoma patients. Since no patients in the thymoma group had a response of Complete or Partial response, the study ended without going to stage two.
Groups:
- Thymoma: Patients classified as having Thymoma. Patients receive 175 mg oral saracatinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Thymic Carcinoma: Patients classified as having Thymic carcinoma. Patients receive 175 mg oral saracatinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Thymoma | Thymic Carcinoma
Started | 12 | 9
Completed | 0 | 0
Not Completed | 12 | 9
Not completed — Disease progression | 9 | 7
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Noncompliance | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thymoma | Thymic Carcinoma | Total
Number analyzed (Participants) | 12 | 9 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 11 | 6 | 17
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (12.25) | 54.2 (17.94) | 51.3 (14.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 5 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 11 | 9 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (Complete and Partial Response)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. The objective response rate will be reported by each disease classification. The percent of patients having an objective response (complete or partial response) will be estimated with a 95% exact binomial confidence interval for the percent of patients receiving drug. Note: there were no objective responses in this trial.
Time Frame: Up to 5 years
Population: All patients with at least one post baseline measurement.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Thymoma | Thymic Carcinoma
Number analyzed (Participants) | 12 | 9
percentage of participants | 0 [0 to 0] | 0 [0 to 0]

2. Secondary Outcome: Progression-free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. This will be examined in an exploratory fashion using Kaplan-Meier estimates. Time until progression, death or last evaluation will be calculated. If a patient did not progress or die, they will be censored at their last evaluation in the analysis.
Time Frame: Time from the date of registration to the first reported outcome event, assessed up to 5 years
Population: All patients who enrolled and received treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Thymoma | Thymic Carcinoma
Number analyzed (Participants) | 12 | 9
months | 5.30 [1.74 to 7.80] | 0.89 [0.86 to 3.95]

3. Secondary Outcome: Overall Survival
Description: Will be examined in an exploratory fashion using Kaplan-Meier estimates. Time until death or last evaluation will be calculated. If a patient did not die, they will be censored in the analysis.
Time Frame: Time from the date of registration to last reported date of survival, assessed up to 5 years
Population: All patients who enrolled and received treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Thymoma | Thymic Carcinoma
Number analyzed (Participants) | 12 | 9
months | 37.47 [12.27 to NA] — The upper confidence interval is not estimable for overall survival in this group due to insufficient number of participants with events. | 6.68 [2.47 to 14.97]

4. Secondary Outcome: Disease Control Rate
Description: Will be examined in an exploratory fashion using Kaplan-Meier estimates. Disease control rate defined as complete response (CR) + partial response (PR) + stable disease (SD). The length of time until progression or until last evaluation will be calculated. For patients who did not progress, they will be censored in the analysis.
Time Frame: Up to 5 years
Population: All patients who enrolled and received treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Thymoma | Thymic Carcinoma
Number analyzed (Participants) | 12 | 9
months | 5.72 [1.84 to 7.80] | 3.55 [NA to NA] — The upper and lower confidence intervals could not be estimated for this group due to insufficient number of participants with events.

5. Secondary Outcome: Expected Toxicities Including Skin Rashes and Diarrhea
Description: Number of patients who had toxicities classified as skin rashes and diarrhea within the adverse events.
Time Frame: Up to 5 years
Population: All patients
Measure: Number; unit: participants
Arm/Group | Thymoma | Thymic Carcinoma
Number analyzed (Participants) | 12 | 9
participants | 10 | 3

ADVERSE EVENTS:
Time Frame: Beginning of treatment until the end of the study, up to 5 years
Arm/Group | Thymoma | Thymic Carcinoma
Serious Adverse Events (participants affected / at risk) | 2/12 | 1/9
Other Adverse Events (participants affected / at risk) | 12/12 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thymoma (N=12) | Thymic Carcinoma (N=9)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0)
Unexpected Change in HEMOGLOBIN level (Investigations) | 1 (1) | 0 (0)
ALBUMIN, SERUM-LOW (HYPOALBUMINEMIA) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PLEURAL EFFUSION (NON-MALIGNANT) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CNS CEREBROVASCULAR ISCHEMIA (Vascular disorders) | 1 (1) | 0 (0)
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 1 (1) | 0 (0)
VESSEL INJURY-VEIN - SVC (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thymoma (N=12) | Thymic Carcinoma (N=9)
BLOOD/BONE MARROW (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
HEMOLYSIS (E.G., IMMUNE HEMOLYTIC ANEMIA, DRUG-RELATED HEMOLYSIS) (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
LEUKOCYTES (TOTAL WBC) (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
LYMPHOPENIA (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
MYOCARDITIS (Cardiac disorders) | 1 (1) | 0 (0)
PALPITATIONS (Cardiac disorders) | 0 (0) | 1 (1)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA - SINUS TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
COGNITIVE DISTURBANCE (Nervous system disorders) | 1 (1) | 0 (0)
OCULAR/VISUAL (Eye disorders) | 1 (1) | 0 (0)
VISION-BLURRED VISION (Eye disorders) | 1 (1) | 0 (0)
ASCITES (NON-MALIGNANT) (Gastrointestinal disorders) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 4 (4) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 6 (6) | 3 (3)
DISTENSION/BLOATING, ABDOMINAL (Gastrointestinal disorders) | 0 (0) | 1 (1)
DYSPHAGIA (DIFFICULTY SWALLOWING) (Gastrointestinal disorders) | 0 (0) | 1 (1)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRITIS (INCLUDING BILE REFLUX GASTRITIS) (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL - OTHER (Gastrointestinal disorders) | 0 (0) | 1 (1)
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 4 (4) | 0 (0)
HEMORRHAGE, GI - ANUS (Gastrointestinal disorders) | 0 (0) | 1 (1)
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) - ORAL CAVITY (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 11 (11) | 3 (3)
PAIN - ABDOMEN NOS (Gastrointestinal disorders) | 4 (4) | 1 (1)
TASTE ALTERATION (DYSGEUSIA) (Gastrointestinal disorders) | 3 (3) | 0 (0)
VOMITING (Gastrointestinal disorders) | 6 (6) | 1 (1)
CONSTITUTIONAL SYMPTOMS - OTHER (General disorders) | 1 (1) | 2 (2)
DYSPNEA (SHORTNESS OF BREATH) (General disorders) | 1 (1) | 1 (1)
EDEMA: HEAD AND NECK (General disorders) | 1 (1) | 0 (0)
EDEMA: LIMB (General disorders) | 2 (2) | 1 (1)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 9 (9) | 7 (7)
FEBRILE NEUTROPENIA (FEVER OF UNKNOWN ORIGIN) (General disorders) | 3 (3) | 1 (1)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 1 (1) | 1 (1)
PAIN - CHEST/THORAX NOS (General disorders) | 4 (4) | 2 (2)
PAIN - OTHER (General disorders) | 0 (0) | 2 (2)
RIGORS/CHILLS (General disorders) | 3 (3) | 0 (0)
SWEATING (DIAPHORESIS) (General disorders) | 1 (1) | 0 (0)
INFECTION - OTHER (Infections and infestations) | 1 (1) | 0 (0)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - ORAL CAVITY-GUMS (GINGIVITIS) (Infections and infestations) | 1 (1) | 0 (0)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - UPPER AIRWAY NOS (Infections and infestations) | 1 (1) | 0 (0)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - URINARY TRACT NOS (Infections and infestations) | 1 (1) | 0 (0)
INFECTION WITH UNKNOWN ANC - LUNG (PNEUMONIA) (Infections and infestations) | 1 (1) | 1 (1)
INFECTION WITH UNKNOWN ANC - ORAL CAVITY-GUMS (GINGIVITIS) (Infections and infestations) | 1 (1) | 0 (0)
INFECTION WITH UNKNOWN ANC - URINARY TRACT NOS (Infections and infestations) | 1 (1) | 0 (0)
ALKALINE PHOSPHATASE (Investigations) | 2 (2) | 3 (3)
ALT, SGPT (SERUM GLUTAMIC PYRUVIC TRANSAMINASE) (Investigations) | 2 (2) | 1 (1)
AST, SGOT(SERUM GLUTAMIC OXALOACETIC TRANSAMINASE) (Investigations) | 3 (3) | 2 (2)
BICARBONATE, SERUM-LOW (Investigations) | 1 (1) | 0 (0)
CREATININE (Investigations) | 1 (1) | 1 (1)
HEMOGLOBIN (Investigations) | 3 (3) | 1 (1)
MUCOSITIS/STOMATITIS (CLINICAL EXAM) - TRACHEA (Investigations) | 1 (1) | 0 (0)
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Investigations) | 0 (0) | 1 (1)
WEIGHT LOSS (Investigations) | 2 (2) | 2 (2)
ALBUMIN, SERUM-LOW (HYPOALBUMINEMIA) (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
ANOREXIA (Metabolism and nutrition disorders) | 7 (7) | 4 (4)
CALCIUM, SERUM-LOW (HYPOCALCEMIA) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
MAGNESIUM, SERUM-LOW (HYPOMAGNESEMIA) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
PHOSPHATE, SERUM-LOW (HYPOPHOSPHATEMIA) (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
POTASSIUM, SERUM-LOW (HYPOKALEMIA) (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
SODIUM, SERUM-LOW (HYPONATREMIA) (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
PAIN - BACK (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
PAIN - EXTREMITY-LIMB (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
PAIN - JOINT (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN - MUSCLE (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
DIZZINESS (Nervous system disorders) | 4 (4) | 0 (0)
INSOMNIA (Nervous system disorders) | 1 (1) | 0 (0)
NEUROPATHY: SENSORY (Nervous system disorders) | 1 (1) | 0 (0)
PAIN - HEAD/HEADACHE (Nervous system disorders) | 2 (2) | 1 (1)
SOMNOLENCE/DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1)
SYNCOPE (FAINTING) (Nervous system disorders) | 0 (0) | 1 (1)
INSOMNIA (Psychiatric disorders) | 2 (2) | 0 (0)
MENTAL STATUS (Psychiatric disorders) | 0 (0) | 1 (1)
MOOD ALTERATION - ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0)
MOOD ALTERATION - DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - URINARY TRACT NOS (Renal and urinary disorders) | 1 (1) | 0 (0)
PAIN - URETHRA (Renal and urinary disorders) | 1 (1) | 0 (0)
PROTEINURIA (Renal and urinary disorders) | 3 (3) | 2 (2)
RENAL/GENITOURINARY - OTHER (Renal and urinary disorders) | 1 (1) | 0 (0)
PAIN - BREAST (Reproductive system and breast disorders) | 1 (1) | 0 (0)
PAIN - VAGINA (Reproductive system and breast disorders) | 1 (1) | 0 (0)
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY - RESPIRATORY TRACT NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ALLERGIC RHINITIS (INCLUDING SNEEZING, NASAL STUFFINESS, POSTNASAL DRIP) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
BRONCHOSPASM, WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 2 (2)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5)
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY - LUNG (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY - NOSE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - UPPER AIRWAY NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
NASAL CAVITY/PARANASAL SINUS REACTIONS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PAIN - SINUS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PLEURAL EFFUSION (NON-MALIGNANT) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
PNEUMONITIS/PULMONARY INFILTRATES (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY/UPPER RESPIRATORY - OTHER (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
VOICE CHANGES/DYSARTHRIA (E.G., HOARSENESS, LOSS OR ALTERATION IN VOICE, LARYNGITIS) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HAIR LOSS/ALOPECIA (SCALP OR BODY) (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
RASH: ACNE/ACNEIFORM (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
SWEATING (DIAPHORESIS) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1)
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less